CLINICAL TRIAL: NCT00957840
Title: Intraventricular Hemorrhage and Post Hemorrhagic Ventricular Dilation: Natural Course, Treatment, and Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Joanna Beachy Ph.D., M.D, University of Utah Neonatology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36114
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Intraventricular Hemorrhage; Premature Infants
Keywords: Omaya reservoirs; cerebral oxygenation; VP shunt; IVH; post hemorrhagic ventricular dilation (PVHD)
MeSH Terms: conditions — Premature Birth | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omaya reservoir group- observational (Other): These infants have been identified with severe enough post hemorrhagic ventricular dilation (PHVD) that they require a reservoir placed for serial cerebro-spinal fluid (CSF) removal. There is no randomization, and infants are compared to a baseline. Observational data will be collected to include NIRS and aEEg which will be done twice weekly, and CSF will be analyzed with each reservoir tap for protein biomarkers.
  Interventions: Procedure: NIRS, aEEG, and CSF concentration of biomarkers

INTERVENTIONS:
Procedure: NIRS, aEEG, and CSF concentration of biomarkers — NIRS and aEEg will be done twice weekly, and CSF will be analyzed with each reservoir tap

SUMMARY:
Intraventricular hemorrhage and its resultant post-hemorrhagic hydrocephalus are significant risk factors for the development of neurodevelopmental delays in preterm infants. The purpose of this study is to determine 1) the incidence of progressive post-hemorrhagic ventricular dilatation (PHVD) in infants with severe intraventricular hemorrhage (IVH), 2) the effect of ventricular dilatation on brain status (cerebral oxygenation, electrical activity, and biomarkers of cerebral damage and repair), and 3) if using ventricular measurements, derived from cranial ultrasound to guide removal of cerebral-spinal fluid through an Omaya reservoir, will help resolve ventricular dilatation and decrease the need for ventriculo-peritoneal (VP) shunt insertion. The hypothesis of this research project is that, by using ventricular measurements to guide the frequency of CSF removal, the rate of VP shunt insertion will be decreased in preterm infants with severe IVH and PHVD. The investigators further hypothesize that cerebral injury, as measured by cerebrospinal fluid (CSF) concentration of biomarkers of neuronal and glial damage and inflammation, will decrease over time with resolution of PHVD.

DETAILED DESCRIPTION:
When an infant has severe IVH noted on cranial ultrasound, s(he) will receive weekly ultrasounds to evaluate progression of ventricular dilatation (standard of care). After the infant is enrolled in this study, Near-Infrared Spectroscopy (NIRS) and Amplitude integrated Electroencephalogram (aEEG) will be performed 1-2 times per week. After Omaya reservoir insertion, ventricular dimensions, based on weekly (standard of care) cranial ultrasounds, will determine frequency of CSF removal. NIRS and aEEG will continue 1-2 times per week to coincide with CSF removal. In addition, 1-2 times per week aliquots of CSF will be stored for evaluation of biomarkers. We will evaluate the impact of IVH and PHVD over time on cerebral oxygenation (NIRS) and cortical electrical activity (aEGG) starting at the time of identification of IVH and correlate these measurements to ventricular dimensions. If an Omaya reservoir is required to control PHVD, we will use ventricular dimensions to guide the frequency of CSF removal and continue to evaluate brain status by measuring cerebral oxygenation (NIRS) and cortical electrical activity (aEGG).

ELIGIBILITY:
Inclusion Criteria:

* severe IVH
* receiving weekly head ultrasounds for monitoring

Exclusion Criteria:

* no or minimal IVH

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2009-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Measure cerebral oxygenation using NIRS and background cerebral electrical activity using aEEG starting at the time of identification of severe IVH to better assess impact of IVH, PHVD, and CSF removal on brain status. | 3 years

SECONDARY OUTCOMES:
Use ventricular measurements to guide frequency of CSF removal. | 3 years
Measure concentration of neuroproteins, such as S100B, GFAP, NSE, TGF-ß, and IL-6, in CSF over time and correlate these markers of cellular damage and inflammation with cerebral oxygenation, electrical activity, and need for VP shunt insertion. | 3 years
Compare the sensitivity and reliability of the different measurement techniques used to determine ventricular dimensions | 3 years
Determine the incidence of progressive PHVD in preterm infants with severe IVH. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Beachy, PhD, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States